CLINICAL TRIAL: NCT04402086
Title: Rheumatology Patient Registry and Biorepository
Status: Recruiting | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Rheumatology Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 2000026608; No NIH funding (Other: 12.07.23)
Record Dates: First submitted 2020-05-20; First posted 2020-05-26 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Rheumatic Diseases; Adult Onset Still Disease; Ankylosing Spondylitis; Psoriatic Arthritis; Reactive Arthritis; Antiphospholipid Syndrome; Systemic Lupus Erythematosus; Behcet Disease; Dermatomyositis; Polymyositis; Giant Cell Arteritis; Lyme Disease; Mixed Connective Tissue Disease; Polymyalgia Rheumatica; Rheumatoid Arthritis; Sarcoidosis; Systemic Sclerosis; Scleroderma; Sjogren's Syndrome; Undifferentiated Connective Tissue Diseases
MeSH Terms: conditions — Rheumatic Diseases; Still's Disease, Adult-Onset; Spondylitis, Ankylosing; Arthritis, Psoriatic; Arthritis, Reactive; Antiphospholipid Syndrome; Lupus Erythematosus, Systemic; Behcet Syndrome; Dermatomyositis; Polymyositis; Giant Cell Arteritis; Lyme Disease; Mixed Connective Tissue Disease; Polymyalgia Rheumatica; Arthritis, Rheumatoid; Sarcoidosis; Scleroderma, Systemic; Scleroderma, Diffuse; Sjogren's Syndrome; Undifferentiated Connective Tissue Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Blood, saliva, urine, stool, and tissue/skin biopsies.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Biorepository: Participants with rheumatic diseases who contributed biospecimen samples (blood, saliva, urine, stool, tissue).

SUMMARY:
To facilitate clinical, basic science, and translational research projects involving the study of rheumatic diseases.

DETAILED DESCRIPTION:
A rheumatology biorepository will be created to permit comparative analyses between the rheumatic diseases in order to increase the understanding of disease pathogenesis. Patients seen at Yale clinics diagnosed with rheumatic diseases are invited to participate in this study. These rheumatic diseases include, but are not limited to: adult onset Still's disease, ankylosing spondylitis, psoriatic arthritis, reactive arthritis, antiphospholipid syndrome, systemic lupus erythematosus, Behcet's disease, dermatomyositis, polymyositis, giant cell arteritis and other vasculitides, Lyme's disease, mixed connective tissue disease, polymyalgia rheumatica, rheumatoid arthritis, sarcoidosis, systemic sclerosis (scleroderma), Sjogren's syndrome, and undifferentiated connective tissue disease.

ELIGIBILITY:
Inclusion Criteria for Rheumatology Patients:

* Patients ≥18 years old with a diagnosis of a rheumatic autoimmune disease including, but not limited to: adult onset Still's disease, ankylosing spondylitis, antiphospholipid syndrome, Behcet's disease, dermatomyositis, giant cell arteritis, mixed connective tissue disease, polymyalgia rheumatica, polymyositis, psoriatic arthritis, reactive arthritis, rheumatoid arthritis, sarcoidosis, scleroderma, Sjogren's syndrome, systemic lupus erythematosus, undifferentiated connective tissue disease and vasculitis.
* Receiving clinical care at Yale Rheumatology clinics

Exclusion Criteria for Rheumatology Patients:

* Unable to provide informed consent
* No patients will be excluded based on gender or ethnicity or pregnancy status.
* Women who are currently pregnant will need to wait to donate a skin biopsy until after they deliver.
* Patients allergic to lidocaine or epinephrine or have a history of impaired wound healing will not be able to donate a skin biopsy.

Inclusion Criteria for Healthy Volunteers:

* Age ≥ 18 years old
* No chronic skin conditions
* No diagnosis of a rheumatic autoimmune disease (e.g., lupus, rheumatoid arthritis)
* Normal BMI

Exclusion Criteria for Healthy Volunteers:

* Unable to provide informed consent.
* Currently pregnant or nursing unless the study goal is to study pregnant or nursing woman.
* Allergies to lidocaine or epinephrine (skin biopsies).
* A history of impaired wound healing (skin biopsies).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The biorepository will consist of both new and established patients with a rheumatic autoimmune disease diagnosis who visit a Yale Rheumatology medical facility and agree to participate in this study. The biorepository will also consist of healthy volunteers who agree to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-08-04 (Actual); Primary Completion 2030-06-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
Correlate outcomes and biomarkers of rheumatic diseases | 10 years
  Evaluate clinical data and biospecimens to correlate outcomes and biomarkers of rheumatic diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Monique Hinchcliff, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
No plan at this time.